CLINICAL TRIAL: NCT04896736
Title: Multisite Tissue Oxygenation Guided Perioperative Care to Reduce Composite Complications in Cardiac Surgical Patients: the BOTTOMLINE-CS Trial
Brief Title: Multisite Tissue Oxygenation Guided Perioperative Care in Cardiac Surgery
Acronym: BOTTOMLINECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Tianjin Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021KY-008-01; 000 (Other: CTGTY)
Record Dates: First submitted 2021-04-26; First posted 2021-05-21 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Brain Ischemia Hypoxia; Muscle; Ischemic; Muscle Hypoxia
Keywords: Cerebral Tissue Oxygen Saturation; Muscular Tissue Oxygen Saturation; Cardiac Surgery; Complications; Multisite Tissue Oxygenation Monitoring
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisite tissue oxygenation monitoring-guided care (Experimental): Details are as follows. • Monitoring: SctO2 monitored using two probes placed on left and right forehead. SstO2 monitored using one probe placed over the forearm brachioradialis muscle on the arm not used for non-invasive blood pressure monitoring.
  • Baseline: The first baseline is measured 12-48 hours before surgery, with the patient supine, awake, calm, eyes closed, and breathing room air or oxygen that is equivalent to the home oxygen rate for patients using home oxygen.
  * Goals: Maintain both SctO2 and SstO2 within 90-110% of the baseline level.
  * Trigger of intervention: SctO2/SstO2 outside of the 90-110% baseline range.
  * Diagnosis:
  * Care team: The caregivers providing SctO2/SstO2-guided care will be trained and given the opportunity to use the intervention protocol in at least 20 patients before the formal study.
  * Treatments: Refer to the algorithm to restore SctO2/SstO2 within 90-110% baseline range.
  Interventions: Other: Multisite tissue oxygenation-guided care
- Usual care (Active Comparator): Patients in the control group will be managed by clinical staff according to usual care. Patients in this group will be monitored using the same tissue oximeter used in the intervention group; however, the screen will be covered by an opaque cloth to prohibit the care givers seeing the monitoring data. The same baseline measurements will be performed in patients allocated to the usual care group.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multisite tissue oxygenation-guided care — The following intervention algorithm is intended to be used as a guidance only. We emphasize the different aspects that can cause changes in SctO2/SstO2 in a systematic approach. We avoid recommending a concrete drug and method of dosing for a specific condition.
  Manage tissue perfusion Preload: overall picture including direct observation of the heart, findings of echocardiography, urine output, blood loss, labs results, HR, BP, PPV, SVV, fluid responsiveness (SV increase >/= 10% following 250 ml fluid bolus) Contractility: direct observation of the heart, findings of echocardiography Stroke volume and heart rate: important determinants of CO Systemic vascular resistance: important determinant of BP Regional vascular resistance: important determinant of tissue perfusion along with perfusion pressure Maintain autoregulation: normalize CO2, avoid potent vasodilators
  Manage arterial blood oxygen content
  Manage tissue metabolic activity
  Arms: Multisite tissue oxygenation monitoring-guided care
Other: Usual care — Usual care in this study means the standard perioperative care. Patients who are meant to receive usual care will receive both cerebral and muscular tissue oxygen saturation monitoring; however, the monitor screen will be covered and the monitoring data will not be used to guide clinical care.
  Arms: Usual care

SUMMARY:
The BOTTOMLINE-CS trial is an international, open, single-center, pragmatic, randomised controlled trial to investigate whether multisite tissue oxygen saturation monitoring-guided perioperative care reduces composite complications within 30 days of randomization in off-pump coronary artery bypass grafting.

DETAILED DESCRIPTION:
Short title: BOTTOMLINE-CS trial Methodology: International, open, single-center, pragmatic, randomised controlled trial Research sites: Tianjin Chest Hospital Objectives: To investigate whether multisite tissue oxygen saturation monitoring-guided perioperative care reduces composite complications within 30 days of randomization in off-pump coronary artery bypass grafting Number of patients: 1960 patients (980 per arm, two arms) Inclusion criteria: Patients aged ≥ 60 years undergoing elective off-pump coronary artery bypass grafting Exclusion criteria: Patient refusal, clinician refusal, preoperative requirement of respiratory support (intubation, CPAP or BiPAP, or high-flow oxygen (>10 L/min)), preoperative requirement of external cardiac assist devices, emergent or urgent surgery, patients expected to die within 30 days, current participation in another clinical trial Statistical analysis: Analyses will be performed on a modified intention-to-treat basis including all randomized patients who had undergone the scheduled surgery and had the record of the primary outcome. Summary statistics for each group, treatment effects, 95% confidence intervals, and p values will be presented for primary and secondary outcomes, and process measures. The primary outcome is a composite of complications arising within 30 days from randomization and will be analyzed using a logistic regression model.

Proposed start date: May 1, 2021 (First patient to be recruited) Proposed end date: April 30, 2023 (Last patient to be recruited) Study duration: 48 months (Starting from the first patient recruitment, spanning patient recruitment, data analysis, and manuscript writing and submission)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 60 years scheduled for elective off-pump CABG.

Exclusion Criteria:

* Inability or refusal to provide consent of participation
* Preoperative requirement of respiratory support (intubation, CPAP or BiPAP, or high-flow oxygen (>10 L/min))
* Preoperative requirement of external cardiac assist device
* Urgent or emergent surgery
* Patients expected to die within 30 days of randomization

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1960 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Composite complication | from the day of surgery (i.e., day 0) until postoperative day 30 for a total of 31 days (individual components may vary)
  The primary outcome is a collapsed (one or more) composite of the following complications with a Clavien-Dindo grade II or greater arising within 30 days of randomization (randomization and surgery are performed on the same day). The patient is regarded as having the event of composite complications if any of the following complications occur (i.e., yes); otherwise, the patient is regarded as not having the event of composite complications. The percentage of patients having the event of composite complications will be used in the primary analysis.
  * Brain complications (delirium, cognition decline, stroke);
  * Cardiac complications (non-fatal cardiac arrest, myocardial injury, heart failure, new-onset symptomatic ventricular arrhythmia);
  * Respiratory failure;
  * Renal complications (AKI stages II and III);
  * Infectious complications;
  * Death.

SECONDARY OUTCOMES:
Atrial fibrillation | from the day of surgery until postoperative day 30
  Atrial fibrillation
  A new diagnosis of AF per the current standard.
Postoperative delirium | from postoperative day 1 throughout postoperative day 5
  Postoperative delirium (assessed using CAM-ICU Worksheet for patients in PACU and ICU, or CAM for patients on the floor). The validated Chinese version will be used for assessment.
  Delirium will be formally assessed as early in the morning as practical and early evening for the initial five postoperative days while patients remain hospitalized because this approach will detect nearly all postoperative delirium. Observed daytime delirium will be recorded and considered as an outcome. Delirium will not be evaluated the evening after surgery because confusion might result from residual anesthetic effects.
Postoperative cognitive decline | Assessed before surgery, on postoperative day 5 and 30
  Postoperative cognitive decline (assessed using 30-points MoCA 7.1 version). The validated Chinese version will be used.
  MoCA evaluates multiple cognitive domains including executive function and is widely used. Validated versions of MoCA are available in many languages including Chinese and German. A decrease of ≥2 points is associated with cognitive decline based on formal neuropsychological testing and considered a clinically meaningful reduction.
Length of hospital stay | from the day of surgery (day 0) until hospital discharge or until day 30, whichever occurs first
  Length of hospital stay in days
Perioperative stroke | Stroke will be assessed from the day of surgery throughout postoperative day 30
  Any stroke per current clinical diagnostic criteria arising during surgery or after surgery until postoperative day 30.
Cardiac complications (one component of the primary outcome) | from the day of surgery (i.e., day 0) until postoperative day 30 for a total of 31 days
  Cardiac complications include:
  * non-fatal cardiac arrest (An absence of cardiac rhythm or presence of chaotic rhythm requiring any component of basic or advanced cardiac life support.)
  * myocardial injury (Myocardial injury is defined as any myocardial infarction (i.e., 4th Universal Definition of myocardial infarction32), or any elevated troponin judged to be due to myocardial ischemia (i.e. without evidence of a non-ischemic etiology, e.g. chronic elevation, pulmonary embolism, sepsis, cardioversion, others) that occurred with the first 30 days after surgery.)
  * heart failure (per current standard diagnostic criteria.)
  * new-onset symptomatic ventricular arrhythmia (per current standard diagnostic criteria.)
Respiratory failure (one component of the primary outcome) | from the day of surgery (i.e., day 0) until postoperative day 30 for a total of 31 days
  Respiratory failure is defined as the requirement of respiratory support (intubation, CPAP or BiPAP, or high-flow oxygen (>10 L/min)) for acute respiratory insufficiency for more than 6 hours after surgery.
Renal complications (one component of the primary outcome) | from the postoperative day 1 until postoperative day 7 for a total of 7 days
  Renal complications in this study refers to acute Kidney Injury stages II and III diagnosed using the Kidney Disease Improving Global Guidelines (KDIGO).
Infectious complications (one component of the primary outcome) | from postoperative day 1 until postoperative day 30 for a total of 30 days
  Infectious complications include the following:
  * Surgical site infection (deep surgical site):
  * Surgical site infection (organ/space)
  * Pneumonia
  * Laboratory confirmed bloodstream infection
  * Infection, source uncertain
  * Sepsis Sepsis will be diagnosed per the Third International Consensus Definitions.38,39 The Task Force defines sepsis as a "life-threatening organ dysfunction due to a dysregulated host response to infection." Clinical diagnosis of organ dysfunction requires a two-point increase in the Sequential [Sepsis-related] Organ Failure Assessment (SOFA) score, starting the day after surgery and continuing throughout hospitalization as shown below (adopted from Singer38).

CONTACTS AND LOCATIONS:
Overall Officials: Jiange Han, Principal Investigator — Tianjin Chest Hospital
Locations (1):
- Tianjin Chest Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
The data will only be available to journals for audits or authorities required by law.

REFERENCES:
- [Background] Li G, Tian DD, Wang X, Feng X, Zhang W, Bao J, Wang DX, Ai YQ, Liu Y, Zhang M, Xu M, Mu DL, Zhao X, Dai F, Yang JJ, Che X, Yanez D, Guo X, Meng L; iMODIPONV Research Group. Muscular Tissue Oxygen Saturation and Posthysterectomy Nausea and Vomiting: The iMODIPONV Randomized Controlled Trial. Anesthesiology. 2020 Aug;133(2):318-331. doi: 10.1097/ALN.0000000000003305. PMID 32667155
- [Derived] Han J, Zhai W, Wu Z, Zhang Z, Wang T, Ren M, Liu Z, Sessler DI, Guo Z, Meng L; Bottomline-CS investigation group. Care guided by tissue oxygenation and haemodynamic monitoring in off-pump coronary artery bypass grafting (Bottomline-CS): assessor blind, single centre, randomised controlled trial. BMJ. 2025 Mar 24;388:e082104. doi: 10.1136/bmj-2024-082104. PMID 40127893

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04896736/SAP_001.pdf